CLINICAL TRIAL: NCT03575416
Title: Prevalence of Multi-morbid Frailty in a Cohort of Subjects Undergoing Cancer Related Surgery
Brief Title: Cancer Anesthesia and Frailty
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Other Study IDs: INT 100-18
Record Dates: First submitted 2018-06-21; First posted 2018-07-02 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Cancer; Anesthesia; Fragility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — C Reactive Protein will be measured from blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Subjects undergoing cancer related surgery at the Fondazione IRCCS Istituto Nazionale dei Tumori - Milano will be consecutively recruited. Data regarding presence of co-morbidities, frailty, cancer staging, and inflammatory status (CRP protein measurement) will be collected preoperatively. Intra-operative data collection will comprehend type and duration of surgery, kind of anesthesia, complications. In-hospital mortality will be considered as the primary endpoint, while secondary outcome measures will be duration of hospital stay and admission to intensive care.

DETAILED DESCRIPTION:
A prospective data collection of pre-intra and postoperative variables will be collected in a cohort of subjects undergoing cancer relate surgery at the Fondazione IRCCS Istituto Nazionale dei Tumori, Milano.

BEFORE SURGERY Subjects will be stratified before surgery according to the following three main clusters: 1) Systemic inflammation: baseline levels of C Reactive Protein; 2) Cancer staging: TNM will be taken into account, together with the type of cancer, previous radio or chemo therapy, and planned/performed surgical procedure; 3) Frailty: subjects will be stratified according to their overall status, taking into account elements of frailty. Co-existing diseases such as diabetes, hypertension, cardiac heart failure, acute myocardial infarction, chronic obstructive disease/asthma, kidney or liver disease (past or present) will be considered. Functional status will be assessed by means of ASA, ECOG status and Possum scores. Frailty will be explored using the mFI and G8 score, the WHO scale, and considering age. Absolute BMI and loss of weight will be used to assess malnutrition.

DURING SURGERY Duration and type of surgery, kind of anesthesia and intra-operative complications will be considered.

AFTER SURGERY Hospital mortality, length of stay, and admission to intensive care will be considered as outcome measures. Major complications, such as myocardial infarction, arrhythmia, cardio circulatory arrest, shock, stroke, pulmonary embolism, kidney failure, delirium, pneumonia or SSI will also be considered.

ELIGIBILITY:
Inclusion Criteria: Subjects undergoing cancer related surgery at the Fondazione IRCSS Istituto Nazionale dei Tumori, Milano

Exclusion Criteria: Day case surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective cohort of subjects undergoing cancer related surgery
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2018-09-01 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days

SECONDARY OUTCOMES:
Duration of hospital stay | 30 days
Admission to intensive care. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Franco Valenza, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Locations (1):
- Fondazione IRCSS Istituto Nazionale dei Tumori, Milan, MI, Italy